CLINICAL TRIAL: NCT04135469
Title: Integration of Tax Preparation Into Pediatric Clinics: A Pilot Study
Brief Title: Tax Preparation Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38575
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Financial Stress; Maternal Distress
Keywords: Tax preparation service; Tax filing; Earned Income Tax Credit (EITC); Child tax credit
MeSH Terms: conditions — Financial Stress | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Referral for tax preparation (Active Comparator): Participants will be given contact information on financial services, including all the free tax preparation services in the city, including Boston Medical Center.
  Interventions: Other: Referral for tax preparation services
- BMC tax preparation (Experimental): A navigator will help the participants with using free tax preparation services located at Boston Medical Center or a service located elsewhere in the city.
  Interventions: Other: Referral for tax preparation services; Other: Navigator assisted tax preparation services at BMC

INTERVENTIONS:
Other: Referral for tax preparation services — Printed materials will be provided with contact information for tax preparation services at BMC and other sites in the city.
Other: Navigator assisted tax preparation services at BMC — A study navigator will assist the participant in accessing the BMC located tax preparation services.
  Arms: BMC tax preparation

SUMMARY:
The goal of this study to understand what percentage of families in the pediatric clinic at Boston Medical Center (BMC) currently file taxes and use free tax preparation and would accept and use referral to a free tax preparation service. The investigators specifically want to understand which of two methods of connecting to free tax preparation (referral versus navigated connection) is more effective. Also studied will be the feasibility of using surveys on financial wellness and other health indicators to track participants' health.

These pilot findings will be used to design a larger study that aims to assess whether integrating free tax preparation services into a pediatric clinic can increase tax filing rates and, as a result, the amount of money families receive in tax refunds. Additionally, the investigators hope to understand whether receiving this service impacts parental stress as well as how parents and babies are using the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Guardian of a child 0-5 years
* English, Spanish, or Haitian-Creole -speaking
* Child is a Boston Medical Center pediatric primary care patient

Exclusion Criteria:

* Guardian not present at time of clinic visit
* Have no taxable income for the calendar year
* Not using BMC for pediatric primary care
* Have already filed their taxes for 2020

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Financial well being | 12 months
  The consumer financial protection bureau (cfpb) financial -well-being questionnaire will be used to assess financial stability. It has 5 items with scores from from 0 to 4 where 4 is the response associated with the best financial well being. Total scores can range from 0 to 16. They are interpreted with a table stratifying the participants age as 19-61 and 62+ and higher scores are more favorable.
Tax refund | 12 months
  A copy of the IRS tax return form will be reviewed to extract the total tax refund amount
Tax credits | 12 months
  A copy of the IRS tax return form will be reviewed to extract the Earned Income Tax Credit and Child Tax Credit amounts

SECONDARY OUTCOMES:
Maternal mental health | 12 months
  The Beck depression inventory is a 21 item instrument with options of responses from 0 to 3. Total scores can range from 0 to 63 and are interpreted with this rubric: 1-10, these ups and downs are considered normal; 11-16, mild mood disturbance; 17-20, borderline clinical depression; 21-30, moderate depression; 31-40, severe depression; over 40, extreme depression
Maternal well being | 12 months
  The Flourishing Scale is a 12-item summary measure of well being. Each of the items is self-rated on a a scale of 0 to 10 where 10 is the best possible response related to well being. Total scores can range from 0 to 120. HIgher scores are associated with higher levels of well being.
Parenting skills | 12 months
  The 'Me as a Parent' questionnaire will be used to assess parenting skills. It is a 16 item scale where a parent is asked to rate how strongly they agree or disagree with the statements. Responses range from 1 to 5 with 1- strongly disagree and 5= strongly agree. Total scores range from 16 to 80 and higher scores are associated with stronger parenting skills.
Maternal healthcare utilization | 12 months
  The electronic medical record for the mother/guardian will be reviewed and the total number and types of health care utilized (eg outpatient visits and hospitalizations) will be abstracted.
Child healthcare utilization | 12 months
  The electronic medical record for the child will be reviewed and the total number and types of health care utilized (eg outpatient visits and hospitalizations) will be abstracted.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Marcil, MD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No